Patterns of Antidepressant therapy and Clinical Outcomes among Ischemic Stroke Survivors

NCT02146274

Statistical Analysis Plan

Document Date: May 24, 2017

# **Statistical Analysis Plan**

Working Title: Patterns of Antidepressant therapy and Clinical Outcomes among Ischemic

Primary Objectives ...... 4

**Stroke Survivors** 

**Registry:** PROSPER; GWTG Stroke, CMS

Investigator: Emily O'Brien

Master Statistician: Haolin Xu

Faculty Statistician: Michael Pencina

### **Table of Contents**

| 1<br>c | - | To estimate the patterns of antidepressant (AD) prescription at hospital discharge among a population of non-traindicated stroke patients. | 4 |
|---|---|---|---|
| | าดเ | To estimate the associations between antidepressant use (any vs. none) and outcomes (home time, all-cause rtality, stroke readmissions, cardiovascular readmissions, and depression-related hospitalizations following charge). | 4 |
| 3 | | Repeat analyses for patients with SSRI information (SSRI vs. other AD). | 4 |
| 4<br>w | - | To examine associations between AD and outcomes in subgroups based on age (80/90), sex, race (white/non-ite), NIH stroke scale (<16/≥16), and history of depression | 4 |
| | | o estimate patterns of AD prescription (AD vs none and SSRI vs other AD) at hospital discharge among prospectiv<br>colled PROSPER patients with ischemic stroke discharge | ely |
| | | To examine associations between antidepressant use (any vs.none) and patient reported outcomes following nemic stroke discharge | |
| 7 | 7. 1 | To examine associations between types of antidepressant used (SSRI vs. other AD) and patient reported outcomes | ŝ. |
| II. | S | Study Population | . 4 |
| III. | ١ | /ariables | . 6 |
| 1 | | Primary exposure variable | 6 |
| 2 | | Other variables | 6 |
| 3 | | Outcomes/Endpoints | 7 |
| IV. | A | Analysis Tasks | . 7 |
| 1 | | Objective 1 | 7 |
| | ٦ | Table 1A. Baseline characteristics of GWTG-Stroke-CMS patients by discharge AD use. | 7 |
| | 7 | Fable 1B. Baseline characteristics of GWTG-Stroke-CMS patients by discharge AD type. | 7 |
| | ٦ | Fable 1. Baseline characteristics of GWTG-Stroke-CMS patients* overall and by discharge AD. | 8 |
| 2 | | Objective 2 | 9 |
| | ٦ | Fable 2. AD use and clinical outcomes following ischemic stroke discharge. | 9 |
| | 1 | Table 3. SSRI vs. non-SSRI use and clinical outcomes following ischemic stroke discharge | 9 |
| 2 | | Objective 3 | 10 |

| | Figure X. Cumulative incidence plots for mortality and readmissions by AD types (Yes vs No, and again for SSRI vs | 5 |
|---|---|---|
| | Non-SSRI). | 10 |
| 4. | Objective 4 | 10 |

**Table 5A**. Baseline characteristics of prospectively enrolled PROSPER patients with ischemic stroke discharge by discharge AD use (any vs none)

**Table 5B**. Baseline characteristics of prospectively enrolled PROSPER patients with ischemic stroke discharge by discharge AD type (SSRI vs. other AD)

## 6. Objective 6

Figure 6. Grotta bar showing AD vs no AD use and mRS following ischemic stroke discharge.

Table 6A. EQ-5D-3L distribution by AD use at discharge, 3 month and 6 month

Table 6B. EQ-5D-3L index values

Table 6C. EQ VAS

Table 6D. PHQ-2 Score distribution

Table 6E. PHQ-2 Score

**Table 6F**. Stroke Impact Scale-16

Table 6G. Fatigue Severity Scale

### 6. Objective 7

Figure 7. Grotta bar showing SSRI vs other AD use and mRS following ischemic stroke discharge.

Table 7A. EQ-5D-3L distribution by SSRI vs other AD use at discharge, 3 month and 6 month

Table 7B. EQ-5D-3L index values

Table 7C. EQ VAS

Table 7D. PHQ-2 Score distribution

Table 7E. PHQ-2 Score

Table 7F. Stroke Impact Scale-16

Table 7G. Fatigue Severity Scale

## I. Primary Objectives

- 1. To estimate the patterns of antidepressant (AD) prescription at hospital discharge among a population of non-contraindicated stroke patients.
- 2. To estimate the associations between antidepressant use (any vs. none) and outcomes (home time, all-cause mortality, stroke readmissions, cardiovascular readmissions, and depression-related hospitalizations following discharge).
- 3. Repeat analyses for patients with SSRI information (SSRI vs. other AD).
- 4. To examine associations between AD and outcomes in subgroups based on age (80/90), sex, race (white/non-white), NIH stroke scale (<16/≥16), and history of depression.
- 5. To estimate patterns of AD prescription (AD vs none and SSRI vs other AD) at hospital discharge among prospectively enrolled PROSPER patients with ischemic stroke discharge
- 6. To examine associations between antidepressant use (any vs.none) and patient reported outcomes following ischemic stroke discharge
- 7. To examine associations between types of antidepressant used (SSRI vs. other AD) and patient reported outcomes.

# Study Population <u>N Patients</u> <u>N Sites</u> <u>% Remained</u>

Starting Population: All PROSPER (GWTG-Stroke linked to CMS\*) patients
enrolled in a fully-participating GWTG hospital with a final clinical
diagnosis of acute ischemic stroke in year 2014

#### 2. Exclusions:

| 1) | Patients FFS ineligible | -5,582 | -2 | 94.7% |
|---|---|---|---|---|
| 2) | Patients discharged before April 2014 | -23,467 | -15 | 76.3% |
| 3) | Patients left AMA/discharge disposition UTD/missing | -255 | -0 | 99.7% |
| 4) | Patients transferred out | -1,486 | -4 | 98.0% |
| 5) | In-hospital deaths | -4,148 | -2 | 94.4% |
| 6) | Discharge AD not documented (historic and new) | -31,801 | -383 | 54.2% |
| 7) | Patients with AD contraindications | -8,507 | -7 | 77.4% |
| | | <mark>=29,177</mark> | <mark>=1,023</mark> | |

3. Final Study Population: 29,177 patients from 1,023 hospitals Study period: Apr 1, 2014 – Dec 31, 2014

**Table.** New AD variable by historic AD variable check in the IS study population.

| Antidepressant<br>Medication(s) At | Antidepressant Medication(s) At Discharge (Historic) | | | |
|---|---|---|---|---|
| Discharge (New) | Missing | Missing 1= Yes 2 = No/ND | | Total |
| | 0 | 6075 | 16234 | 22309 |
| . = Missing | 0 | 20.82 | 55.64 | 76.46 |
| IVIISSIIIG | 0 | 27.23 | 72.77 | |
| | 0 | 99.72 | 99.71 | |
| | 1063 | 9 | 0 | 1072 |
| 1 - Vee CCDI | 3.64 | 0.03 | 0 | 3.67 |
| 1 = Yes, SSRI | 99.16 | 0.84 | 0 | |
| | 15.63 | 0.15 | 0 | |

<sup>\*</sup> Linkage to CMS implies that patients are at age of 65 or older, linked with first admission

| Antidepressant<br>Medication(s) At | Antidepressant Medication(s) At Discharge (Historic) | | | |
|---|---|---|---|---|
| Discharge (New) | Missing | 1= Yes | 2 = No/ND | Total |
| | 438 | 8 | 0 | 446 |
| 2 = Yes, any other | 1.50 | 0.03 | 0 | 1.53 |
| antidepressant class | 98.21 | 1.79 | 0 | |
| | 6.44 | 0.13 | 0 | |
| | 5302 | 0 | 48 | 5350 |
| 3 = No/ND | 18.17 | 0 | 0.16 | 18.34 |
| טאו /טאו – 3 | 99.10 | 0 | 0.90 | |
| | 77.94 | 0 | 0.29 | |
| Total | 6803 | 6092 | 16282 | 29177 |
| Total | 23.32 | 20.88 | 55.80 | 100 |

Color code: AD Yes patients, AD No patients

#### II. Variables

#### 1. Primary exposure variable

<u>Any antidepressant prescription at hospital discharge</u> (yes vs. no, derived from a combination of historic and revised antidepressant variables)

- Historic AD variable: AD Yes / AD No

- New AD variable: Yes, SSRI / Yes, other AD class

SSRI (selective serotonin reuptake inhibitors) are defined as any of the following: Citalopram (Celexa), Escitalopram (Lexapro), Fluoxetine (Prozac), Paroxetine (Paxil, Pexeva), Sertraline (Zoloft). Other antidepressant therapy will be defined as all other non-SSRI antidepressants. SSRI analyses will be limited to patients with complete data on the new AD variable.

| AD | Frequency | Percent |
|-------|-----------|---------|
| Yes | 7,593 | 26.02 |
| No | 21,584 | 73.98 |
| Total | 29,177 | 100 |

| SSRI | Frequency | Percent |
|---------------|-----------|---------|
| Yes, SSRI | 1,072 | 70.62 |
| Yes, other AD | 446 | 29.38 |
| Total | 1,518 | 100 |

| Variable | Level | Overall AD YES (N=29177) (N=7593) | | AD NO<br>(N=21584) | | P-value+ | | |
|---|---|---|---|---|---|---|---|---|
| History of depression | Yes<br>No | 4341<br>24836 | 14.88<br>85.12 | 3309<br>4284 | 43.58<br>56.42 | 1032<br>20552 | 4.78<br>95.22 | <.0001 |
| AD prior to admission | Yes<br>No<br>Missing | 6432<br>22437<br>308 | 22.28<br>77.72<br>1.06 | 5678<br>1836<br>79 | 75.57<br>24.43<br>1.04 | 754<br>20601<br>229 | 3.53<br>96.47<br>1.06 | <.0001 |

| Variable | able Level Overall (N=1518) | | SSRI YES<br>(N=1072) | | SSRI NO<br>(N=446) | | P-value+ | |
|---|---|---|---|---|---|---|---|---|
| History of depression | Yes<br>No | 667<br>851 | 43.94<br>56.06 | 474<br>598 | 44.22<br>55.78 | 193<br>253 | 43.27<br>56.73 | 0.7361 |
| AD prior to admission | Yes<br>No<br>Missing | 1125<br>380<br>13 | 74.75<br>25.25<br>0.86 | 800<br>262<br>10 | 75.33<br>24.67<br>0.93 | 325<br>118<br>3 | 73.36<br>26.64<br>0.67 | 0.4238 |

## 2. Other variables

Demographics: Age, race, gender, insurance status, medical history (depression, stroke,

TIA, DM, CAD, AF, HF, HTN, PVD, smoking)

Presentation variables: EMS transport, ambulatory status, initial NIHSS, prior antidepressant use

In-hospital variables: Dysphagia screening, DVT prophylaxis, t-PA, t-PA date/time, VTE

interventions, documented DVT/PE, antithrombotics by day 2

Discharge variables: Discharge disposition, ambulatory status at discharge, ICD-9 discharge

diagnosis, Antiplatelet/anticoagulant/HTN/AD meds, stroke education,

smoking cessation, assessment for rehabilitation services

Hospital variables: Primary stroke center; comprehensive stroke center, teaching status,

hospital bed size, rural location, region, annual volume of IS admissions

#### 3. Outcomes/Endpoints

### Primary:

 Home-time: Total number of days spent alive and outside of a hospital, skilled nursing facility, or inpatient rehabilitation facility since discharge

#### Secondary:

- All-cause mortality: Ascertained on the basis of the death date recorded in the denominator/vital status file.
- All-cause readmission: Readmission date will be ascertained from the inpatient institutional file.
- Stroke/TIA readmission: Readmission date will be ascertained from the inpatient institutional file and determined by ICD-9-CM principal diagnoses code of 430, 431, 432.x-435.x, and 436 on the inpatient claim. Ischemic stroke and hemorrhagic stroke will be analyzed separately.
- Cardiovascular readmission: CV Readmission date will be ascertained from the inpatient institutional file and determined by DRG 104–112, 115–118, 121–145, 479, 514–518, 525–527, 535, 536, and 547–558 on the inpatient claim.
- Non-cardiovascular readmission: All readmissions not meeting CV readmission criteria.
- Depression related readmission: Completed suicide, suicide attempt or major depressive episode (major depressive disorder [296.2, 296.3, 296.5, 298.0, or 311], completed suicide/suicide attempt [E950-E959\*], suicide ideation [V62.84], or suicide tendencies [300.9])

### III. Analysis Tasks

#### 1. Objective 1

Aim: To describe patient and hospital characteristics in the study population by discharge AD.

Analysis: Patient characteristics including demographics, medical history, initial vital signs, lab results and hospital characteristics will be described for the study population by discharge AD use. Categorical variables will be presented as proportions, and continuous variables will be presented as mean (standard deviation). We will compare the respective distributions of baseline characteristics among patients receiving 1) Any AD vs. no AD, and 2) SSRI vs. non-SSRI. Differences between groups will be evaluated using chi-square tests for categorical variables and Kruskal-Wallis tests for continuous variables.

Output: <u>Table 1</u> (patient baseline table)

**Table 1A.** Baseline characteristics of GWTG-Stroke-CMS patients by discharge AD use.

| <u>Variables</u> | AD at Discharge | No AD at Discharge | Standardized differences, % P-value | * |
|---|---|---|---|---|

**Table 1B.** Baseline characteristics of GWTG-Stroke-CMS patients by discharge AD type.

| <u>Variables</u> | SSRI at Discharge | Other AD at Discharge | Standardized differences, % | P-value* |
|---|---|---|---|---|
|---|---|---|---|---|

(Detailed table entries on next page)

<sup>\*</sup>Given the potential for under-capture of completed suicides and suicide attempts, depression-related admission outcomes will be considered exploratory (reference: <a href="http://www.mini-sentinel.org/work">http://www.mini-sentinel.org/work</a> products/HealthOutcomes/MS HOI SuicideReport.pdf)

Table 1 Baseline characteristics of GWTG-Stroke-CMS natients\* overall and by discharge AD

| <u>Variables</u> | AD at Discharge | No AD at Discharge | StdDiff, % | P-value* |
|---|---|---|---|---|
| Demographics | | | | |
| Age, year, mean (SD) | | | | |
| Gender: Female | | | | |
| Race/Ethnicity | | | | |
| Medical History | | | | |
| Depression | | | | |
| Atrial Fibrillation | | | | |
| Stroke/TIA | | | | |
| CAD/MI | | | | |
| Carotid Stenosis | | | | |
| Diabetes Mellitus | | | | |
| PVD | | | | |
| Hypertension | | | | |
| Smoker | | | | |
| Dyslipidemia | | | | |
| Heart Failure | | | | |
| Medications prior to admission | | | | |
| Antidepressants | | | | |
| Anti-hypertensives | | | | |
| Cholesterol-reducers | | | | |
| Diabetic medications | | | | |
| Presentation | | | | |
| EMS transport | | | | |
| Initial NIHSS | | | | |
| Onset to arrival times (Prehospital delay) | | | | |
| <2 hours | | | | |
| 2-4 hours | | | | |
| >4 hours | | | | |
| Symptoms resolved at time of presentation | | | | |
| Ambulatory status on admission | | | | |
| Labs | | | | |
| Body Mass Index, mean (SD) | | | | |
| Systolic blood pressure, mean (SD) | | | | |
| Hemoglobin A1C, mean (SD) | | | | |

Hemoglobin A1C, mean (SD) LDL-C, mean (SD)

# **Hospital characteristics**

Teaching status **Rural location** Region **Primary Stroke Centers** Comprehensive Stroke Centers Hospital size, mean (SD) Annual IS admission volume, mean (SD)

All numbers presented are proportions of patient in the study population, unless specified otherwise.

Page 8 of 21

<sup>\*</sup> P-values from chi-squared tests for independence for categorical variables and Wilcoxon rank sum tests for continuous variables

**Aim:** To estimate the associations between antidepressant use (any vs. none) and outcomes (home time, all-cause mortality, all-cause readmission recurrent stroke [ischemic, hemorrhagic], cardiovascular rehospitalization, and depression-related hospitalization [suicidality or major depressive episode] following discharge).

Analysis: Because patients who receive AD may differ from those who do not on important baseline and clinical characteristics that may affect the likelihood of adverse events, we will use inverse probability of treatment weighting (IPW) when assessing treatment effects. IPT weighting will be accomplished in two steps: First, we will use a logistic regression model to assign a probability of treatment selection to each patient based on the distribution of a defined set of covariates (listed above). The binary outcome for the selection model will be AD treatment (Y/N). In the second step, we will weight subject by the inverse of this assigned treatment probability, resulting in a pseudorandomization of patients to AD vs. no AD treatment. The distribution of baseline patient characteristics for each treatment group will be assessed after weighting to determine adequacy of the selection model.

Following IPW, we will compare primary and secondary endpoints between treatment groups. Unadjusted rates of all-cause mortality, all-cause readmission, CV readmission, depression-related admission and stroke/TIA readmission will be examined using a Cox proportional hazards model with AD use as the single independent variable. Adjusted event rates will then be estimated using the same model with IPW included for each subject. Within-hospital clustering will be accounted for using robust estimator approach.

Home time will be examined first as a continuous variable in a linear regression model and then as a dichotomous outcome in an IPW-weighted logistic regression model, using 100% of time spent at home over 1 year as the primary outcome of interest.

Methods will be repeated for SSRI vs. non-SSRI with corresponding modeling of clinical outcomes.

Output: Table 2 (AD vs No AD), Table 3 (SSRI vs not SSRI)

**Table 2.** AD use and clinical outcomes following ischemic stroke discharge.

| Outcomes | AD | No AD<br>(ref) | Unadjusted HR<br>(95% CI) | Adjusted HR<br>(95% CI) | P-value |
|---|---|---|---|---|---|
| <b>Table 3.</b> SSRI vs | . non-SSRI use and | d clinical outco | omes following ischem | ic stroke discharge. | |
| Outcomes | SSRI | Other AD<br>(ref) | Unadjusted HR<br>(95% CI) | Adjusted HR<br>(95% CI) | P-value |

Home time: 100% (OR)
All-cause mortality
Readmission

All-cause
Cardiovascular
Stroke/TIA
Ischemic Stroke
Hemorrhagic Stroke
Depression-related readmission

Unadjusted Difference
(95% CI)

Home time days, mean (SD)

Version 2 Last update05/24/2017

#### 3. Objective 3

**Aim:** To describe 1y mortality and readmission outcomes by plotting the cumulative incidence functions.

**Analysis:** We will limit the population to <u>patients naïve to AD</u> on admission and construct Kaplan-Meier curves for all-cause mortality at 1 year following the index hospitalization for patients prescribed AD at hospital discharge. Log-rank tests will be used to examine mortality differences between AD treatment groups.

For the other non-mortality endpoints, we will calculate incidence at 1 year based on estimates from the cumulative incidence function, to account for the competing risk of mortality. Gray tests will be used to test for differences between groups for these outcomes.

We will then restrict the study population to patients receiving AD at hospital discharge and analyses will be repeated for SSRI vs. non-SSRI antidepressants.



**Figure X.** Cumulative incidence plots for mortality and readmissions by AD types (Yes vs No, and again for SSRI vs Non-SSRI).

#### 4. Objective 4

Aim: Perform subgroup analyses.

Analysis: Because AD use and outcomes may vary by patient characteristics, we will repeat modeling of these associations by the following subgroups: Age (65-80, 80-90, 90+), sex (male vs. female), race (white vs. non-white), NIH stroke scale (<16 vs.  $\ge16$ ), and medical history of depression.

Repeat Tables 2 and 3 in subgroups defined.

## 5. Objective 5

**Aim:** To describe baseline patient and hospital characteristics in the prospectively enrolled PROSPER study population with ischemic stroke discharge by discharge antidepressant use (any vs none).

**Analysis:** Patient characteristics including demographics, medical history, initial vital signs, lab results and hospital characteristics will be described for the study population by discharge AD use (any vs

none). Categorical variables will be presented as proportions, and continuous variables will be presented as mean (standard deviation). We will compare the respective distributions of baseline characteristics among patients receiving any AD vs. none. Differences between groups will be evaluated using chi-square tests for categorical variables and Kruskal-Wallis tests for continuous variables.

**Output:** Table 5A. (patient baseline table)

Table 5A. Baseline characteristics of prospectively enrolled PROSPER patients with ischemic stroke

| <u>Variables</u> | AD at Discharge | No AD at Discharge | StdDiff, % | P-value* |
|---|---|---|---|---|
| Demographics | | | | |
| Age, year, mean (SD) | | | | |
| Gender: Female | | | | |
| Race/Ethnicity | | | | |
| Medical History | | | | |
| Depression | | | | |
| Atrial Fibrillation | | | | |
| Stroke/TIA | | | | |
| CAD/MI | | | | |
| Carotid Stenosis | | | | |
| Diabetes Mellitus | | | | |
| PVD | | | | |
| Hypertension | | | | |
| Smoker | | | | |
| Dyslipidemia | | | | |
| Heart Failure | | | | |
| Medications prior to admission | | | | |
| Antidepressants | | | | |
| Anti-hypertensives | | | | |
| Cholesterol-reducers | | | | |
| Diabetic medications | | | | |
| Presentation | | | | |
| FMS transport | | | | |

EMS transport

Initial NIHSS

Onset to arrival times (Prehospital delay)

<2 hours

2-4 hours

>4 hours

Symptoms resolved at time of presentation

Ambulatory status on admission

#### Labs

Body Mass Index, mean (SD) Systolic blood pressure, mean (SD) Hemoglobin A1C, mean (SD)

LDL-C, mean (SD)

#### **Hospital characteristics**

Teaching status

**Rural location** 

Region

**Primary Stroke Centers** 

**Comprehensive Stroke Centers** 

Hospital size, mean (SD)

Annual IS admission volume, mean (SD)

All numbers presented are proportions of patient in the study population, unless specified otherwise.

\* P-values from chi-squared tests for independence for categorical variables and Wilcoxon rank sum tests for continuous variables

**Table 5B.** Baseline characteristics of prospectively enrolled PROSPER patients with ischemic stroke discharge by discharge AD type.

| <u>Variables</u> | SSRI at Discharge | Other AD at<br>Discharge | StdDiff, % | P-value* |
|---|---|---|---|---|
| Demographics | | | | |
| Age, year, mean (SD) | | | | |
| Gender: Female | | | | |
| Race/Ethnicity | | | | |
| Medical History | | | | |
| Depression | | | | |
| Atrial Fibrillation | | | | |
| Stroke/TIA | | | | |
| CAD/MI | | | | |
| Carotid Stenosis | | | | |
| Diabetes Mellitus | | | | |
| PVD | | | | |
| Hypertension | | | | |
| Smoker | | | | |
| Dyslipidemia | | | | |
| Heart Failure | | | | |
| Medications prior to admission | | | | |
| Antidepressants | | | | |
| Anti-hypertensives | | | | |
| Cholesterol-reducers | | | | |
| Diabetic medications | | | | |
| Presentation | | | | |
| EMS transport | | | | |
| Initial NIHSS | | | | |
| Onset to arrival times (Prehospital delay) | | | | |
| <2 hours | | | | |
| 2-4 hours | | | | |
| >4 hours | | | | |
| Symptoms resolved at time of presentatio | n | | | |
| Ambulatory status on admission | | | | |
| Labs | | | | |
| Body Mass Index, mean (SD) | | | | |
| Systolic blood pressure, mean (SD) | | | | |
| Hemoglobin A1C, mean (SD) | | | | |

#### **Hospital characteristics**

LDL-C, mean (SD)

Teaching status
Rural location
Region
Primary Stroke Centers
Comprehensive Stroke Centers
Hospital size, mean (SD)

Annual IS admission volume, mean (SD)

**Aim:** To estimate the associations between antidepressant use (any vs. none) and patient reported outcomes (modified Rankin Scale, EQ-5D-3L Health Profile, PHQ-2 score, SIS-16 score and Fatigue Severity Scale score).

**Figure 6.** Grotta bar showing AD vs no AD use and mRS following ischemic stroke discharge.



## EQ-5D-3L Health Profile

Table 6A. EQ-5D-3L distribution by AD use at discharge, 3 month and 6 month

| EQ-5D-3L Din | nension | AD | (% Subjec | ts) | Not on AD (% Subjects) | | |
|---|---|---|---|---|---|---|---|
| | | At | 3 | 6 | At | 3 | 6 |
| | | discharge | month | month | discharge | month | month |
| Mobility | Level 1 | | | | | | |
| | Level 2 | | | | | | |
| | Level 3 | | | | | | |
| Self-Care | Level 1 | | | | | | |
| | Level 2 | | | | | | |
| | Level 3 | | | | | | |
| Usual Activity | Level 1 | | | | | | |
| | Level 2 | | | | | | |

| | Level 3 |
|--------------------|---------|
| Pain/Discomfort | Level 1 |
| | Level 2 |
| | Level 3 |
| Anxiety/Depression | Level 1 |
| | Level 2 |
| | Level 3 |

PROSPER

# Table 6B. EQ-5D-3L index values

| EQ-5D-3L index value | AD | | | Not on AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |

# Table 6C. EQ VAS

| EQ VAS | AD | | | Not on AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |

# Table 6D. PHQ-2 Score distribution

| PHQ-2 Score | AD (% Subjects) | | | Not on AD (% Subjects) | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |
| 5 | | | | | | |
| 6 | | | | | | |

# Table 6E. PHQ-2 Score

| PHQ-2 Score | AD | | | Not on AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |
| % Subjects >= 3 | | | | | | |

Table 6F. Stroke Impact Scale-16

| SIS-16 | AD | | | Not on AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 – 75 percentile) | | | | | | |
| Percent at floor (SIS16 = 0) | | | | | | |
| Percent at Ceiling (SIS16 = 100) | | | | | | |

# Table 6G. Fatigue Severity Scale

| Fatigue Severity Scale | AD | | | Not on AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |
| % Subjects >= 36 | | | | | | |

**Aim:** To estimate the associations between antidepressant use (SSRI vs. other) and patient reported outcomes (modified Rankin Scale, EQ-5D-3L Health Profile, PHQ-2 score, SIS-16 score and Fatigue Severity Scale score).

**Figure 7.** Grotta bar showing SSRI vs other AD use and mRS following ischemic stroke discharge.



### EQ-5D-3L Health Profile

Table 7A. EQ-5D-3L distribution by AD type use at discharge, 3 month and 6 month

| EQ-5D-3L Di | mension | SSRI | (% Subjec | ts) | Other type AD (% Subjects) | | |
|---|---|---|---|---|---|---|---|
| | | At | 3 | 6 | At | 3 | 6 |
| | | discharge | month | month | discharge | month | month |
| Mobility | Level 1 | | | | | | |
| | Level 2 | | | | | | |
| | Level 3 | | | | | | |
| Self-Care | Level 1 | | | | | | |
| | Level 2 | | | | | | |
| | Level 3 | | | | | | |
| Usual Activity | Level 1 | | | | | | |
| | Level 2 | | | | | | |
| | Level 3 | | | | | | |
| Pain/Discomfort | Level 1 | | | | | | |

| | Level 2 |
|--------------------|---------|
| | Level 3 |
| Anxiety/Depression | Level 1 |
| | Level 2 |
| | Level 3 |

PROSPER

# Table 7B. EQ-5D-3L index values

| EQ-5D-3L index value | | SSRI | | ( | Other AD | .D |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |

# Table 7C. EQ VAS

| EQ VAS | SSRI | | | ( | Other AD | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |

# Table 7D. PHQ-2 Score distribution

| PHQ-2 Score | SSRI (% Subjects) | | | Other A | D (% Subj | ects) |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |
| 5 | | | | | | |
| 6 | | | | | | |

# Table 7E. PHQ-2 Score

| PHQ-2 Score | SSRI | | | ( | Other AD | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |
| % Subjects >= 3 | | | | | | |

| SIS-16 | SSRI | | ( | Other AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 – 75 percentile) | | | | | | |
| Percent at floor (SIS16 = 0) | | | | | | |
| Percent at Ceiling (SIS16 = 100) | | | | | | |

# Table 7G. Fatigue Severity Scale

| Fatigue Severity Scale | SSRI | | ( | Other AD | | |
|---|---|---|---|---|---|---|
| | At | 3 | 6 | At | 3 | 6 |
| | discharge | month | month | discharge | month | month |
| Mean (Standard error) | | | | | | |
| Median (25 <sup>th</sup> – 75 <sup>th</sup> percentile) | | | | | | |
| % Subjects >= 36 | | | | | | |